CLINICAL TRIAL: NCT03987919
Title: A Phase 3, Randomized, Open-Label Trial Comparing Efficacy and Safety of Tirzepatide Versus Semaglutide Once Weekly as Add-on Therapy to Metformin in Patients With Type 2 Diabetes
Brief Title: A Study of Tirzepatide (LY3298176) Versus Semaglutide Once Weekly as Add-on Therapy to Metformin in Participants With Type 2 Diabetes
Acronym: SURPASS-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17001; I8F-MC-GPGL (Other: Eli Lilly and Company); 2018-004422-29 (EudraCT Number)
Record Dates: First submitted 2019-06-14; First posted 2019-06-17 (Actual); Results first posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2021-07

CONDITIONS: Type 2 Diabetes
Keywords: T2DM; GLP-1 RA; Glucose-dependent insulinotropic polypeptide (GIP); glucagon-like peptide-1 (GLP-1); GIP/GLP-1 dual receptor agonist
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide; semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 5 mg Tirzepatide (Experimental): 5 milligrams (mg) tirzepatide administered subcutaneously (SC) once a week.
  Interventions: Drug: Tirzepatide
- 10 mg Tirzepatide (Experimental): 10 mg tirzepatide administered SC once a week.
  Interventions: Drug: Tirzepatide
- 15 mg Tirzepatide (Experimental): 15 mg tirzepatide administered SC once a week.
  Interventions: Drug: Tirzepatide
- 1 mg Semaglutide (Active Comparator): 1 mg semaglutide administered SC once a week.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 10 mg Tirzepatide; 15 mg Tirzepatide; 5 mg Tirzepatide
Drug: Semaglutide — Administered SC
  Arms: 1 mg Semaglutide

SUMMARY:
The reason for this study is to compare the effect of the study drug tirzepatide to semaglutide on blood sugar levels in participants with type 2 diabetes. The study will last approximately 47 weeks and may include about 12 visits.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with type 2 diabetes mellitus (T2DM)
* Have HbA1c between ≥7.0% and ≤10.5%
* Be on stable treatment with unchanged dose of metformin >1500 mg/day for at least 3 months prior to screening
* Be of stable weight (±5%) for at least 3 months before screening
* Have a body mass index (BMI) ≥25 kilograms per meter squared (kg/m²) at screening

Exclusion Criteria:

* Have type 1 diabetes mellitus
* Have had chronic or acute pancreatitis any time prior to study entry
* Have proliferative diabetic retinopathy or diabetic maculopathy or nonproliferative diabetic retinopathy requiring acute treatment
* Have disorders associated with slowed emptying of the stomach, or have had any stomach surgeries for the purpose of weight loss
* Have acute or chronic hepatitis, signs and symptoms of any other liver disease, or blood alanine transaminase (ALT) enzyme level >3.0 times the upper limit of normal (ULN) for the reference range, as determined by the central laboratory. Participants with nonalcoholic fatty liver disease (NAFLD) are eligible for participation in this trial only if there ALT level is ≤3.0 the ULN for the reference range
* Have an estimated glomerular filtration rate <45 milliliters/minute/1.73 m² (or lower than the country specific threshold for using the protocol required dose of metformin per local label)
* Have had a heart attack, stroke, or hospitalization for congestive heart failure in the past 2 months
* Have a personal or family history of medullary thyroid carcinoma or personal history of multiple endocrine neoplasia syndrome type 2
* Have been taking any other diabetes medicines other than metformin during the last 3 months
* Have been taking weight loss drugs, including over-the-counter medications during the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1879 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (127):
- United States (51):
  - Cahaba Research, Birmingham, Alabama
  - Syed Research Consultants Llc, Sheffield, Alabama
  - National Research Institute - Huntington Park, Huntington Park, California
  - Catalina Research Institute, LLC, Montclair, California
  - Valley Clinical Trials, Inc., Northridge, California
  - National Research Institute - Huntington Park, Panorama City, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - University Clinical Investigators, Inc., Tustin, California
  - CMR of Greater New Haven, Hamden, Connecticut
  - Clinical Research of South Florida, Coral Gables, Florida
  - East Coast Institute for Research at The Jones Center, Lake City, Florida
  - South Florida Clinical Research Institute, Margate, Florida
  - Suncoast Research Group, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Oviedo Medical Research, Oviedo, Florida
  - South Broward Research, Pembroke Pines, Florida
  - United Osteoporosis Center, Gainesville, Georgia
  - Sky Clinical Research Network, Union City, Georgia
  - Elite Clinical Trials, Blackfoot, Idaho
  - University of Iowa Hospital & Clinic, Iowa City, Iowa
  - Cotton O'Neil Clinic, Topeka, Kansas
  - Cotton O'Neil Diabetes and Endocrinology Center, Topeka, Kansas
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Clinvest Research LLC, Springfield, Missouri
  - Premier Research, Trenton, New Jersey
  - Albany Medical College, Division of Community Endocrinology, Albany, New York
  - PharmQuest, Greensboro, North Carolina
  - Diabetes & Endocrinology Consultants, PC, Morehead City, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Aventiv Research Inc, Columbus, Ohio
  - Intend Research, LLC, Norman, Oklahoma
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Detweiler Family Medicine & Associates, Lansdale, Pennsylvania
  - Green & Seidner Family Practice Associates, Lansdale, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Preferred Clinical Research-St. Clair, Pittsburgh, Pennsylvania
  - Holston Medical Group, Bristol, Tennessee
  - Dallas Diabetes Research Center, Dallas, Texas
  - Biopharma Informatic, Inc., Houston, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Carl R. Meisner Medical Clinic, PLLC, Sugar Land, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - Burke Internal Medicine and Research, Burke, Virginia
  - Capital Clinical Research Center, Olympia, Washington
  - The Vancouver Clinic, Vancouver, Washington
- Argentina (13):
  - CEDIC, CABA, AR-B
  - CIPREC, Ciudad Autonoma de Buenos Aire, AR-B
  - Investigaciones Medicas Imoba Srl, Buenos Aires, AR-C
  - CEMEDIAB, C.a.b.a., AR-C
  - Sanatorio Norte, Santiago del Estero, AR-G
  - Centro de Investigaciones Metabólicas (CINME), CABA, Buenos Aires
  - Centro Médico Viamonte, CABA, Buenos Aires
  - Centro Medico Dr Laura Maffei Investigacion Clinica Aplicada, CABA, Buenos Aires
  - Mautalen Salud e Investigacion-Centro de Osteopatías Médicas, Ciudad Autonoma de Buenos Air, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata, Buenos Aires
  - CIPADI, Godoy Cruz, Mendoza Province
  - Instituto Centenario, Ciudad Autonoma de Buenos Aire
  - Cent Priva Especiali Médicas Ambulatorias Inve Clin CEMAIC, Córdoba
- Australia (13):
  - Paratus Clinical Research Western Sydney, Blacktown, Au-nsw
  - Campbelltown Medical & Dental Centre, Campbelltown, Au-nsw
  - Paratus Clinical Research Central Coast, Kanwal, Au-nsw
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - GenesisCare - Bundaberg, Bundaberg, Queensland
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - Core Research Group, Milton, Queensland
  - AusTrials, Taringa, Queensland
  - Eastern Clinical Research Unit, Box Hill, Victoria
  - Barwon Health - The Geelong Hospital, Geelong, Victoria
  - GenesisCare - Wexford Medical Centre WA, Joondalup, Western Australia
  - GenesisCare - Wexford Medical Centre WA, Murdoch, Western Australia
  - Adelaide Medical Solutions, Woodville South
- Brazil (7):
  - CEDOES, Vitória, Br-es
  - ISPEM - Instituto São José dos Campos em Pesquisas Médicas, São José dos Campos, Br-sp
  - CPQuali Pesquisa Clínica, São Paulo, Br-sp
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo, Br-sp
  - Centro de Pesquisas em Diabetes, Porto Alegre, Rio Grande do Sul
  - CPCLIN, São Paulo, São Paulo
  - Dr. Consulta Clínica Médica LTDA, São Paulo
- Canada (8):
  - Milestone Research Inc., London, Ca-on
  - Bluewater Clinical Research Group Inc., Sarnia, Ca-on
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto, Ca-on
  - Manna Research, Lévis, Ca-qc
  - Manna Research - Burlington North, Burlington, Ontario
  - Manna Research - Burlington North, Nepean, Ontario
  - Manna Research - Burlington North, Stoney Creek, Ontario
  - Manna Research - Burlington North, Toronto, Ontario
- Israel (9):
  - Meir Medical Center, Kfar Saba, Central District
  - Clalit Health Services - Shuali Clinic, Raanana, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Diabetes Medical Center, Tel Aviv, Il-ta
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Clalit Health Services - Sakhnin Community Clinic, Sakhnin
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Rambam Health Care Campus, Haifa, Ḥeifā
  - Linn Medical Center, Haifa, Ḥeifā
- Mexico (8):
  - Centro Especializado en Diabetes Obesidad y Enfermedades, México, D.F.
  - Diseno y Planeacion en Investigacion Medica, Guadalajara, Jalisco
  - Instituto Jalisciense de Investigacion en Diabetes y Obesida, Guadalajara, Jalisco
  - Unidad de Investigaci�n Cl�nica Cardiometabolica de Occidente, Guadalajara, Mx-jal
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, N.L.
  - Unidad Médica para la Salud Integral, San Nicolás de los Garza, Nuevo León
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, Ciudad Madero, Tamaulipas
  - Investigacion en Salud y Metabolismo S.C, Chihuahua City
- Puerto Rico (4):
  - Paola Mansilla-Letelier, MD, Guaynabo, PR
  - Research and Cardiovascular Corp., Ponce, PR
  - Martha Gomez Cuellar M.D., San Juan, PR
  - Clinical Research Puerto Rico, San Juan
- United Kingdom (14):
  - Oldfield Surgery, Bath, Avon
  - Staploe Medical Centre, Ely, Gb-cam
  - Fowey River Practice, Fowey, Gb-con
  - Oak Tree Surgery, Liskeard, Gb-con
  - Rame Medical Ltd, Torpoint, Gb-con
  - Royal Primary Care Chesterfield North west, Chesterfield, Gb-dby
  - Knowle House Surgery, Plymouth, Gb-dev
  - Queen Alexandra Hospital, Portsmouth, Gb-ham
  - Lister Hospital, Stevenage, Gb-hrt
  - Oakenhurst Medical Practice, Blackburn, Gb-lan
  - Rowden Surgery, Chippenham, Gb-wil
  - Leicester General Hospital, Leicester, Leicestershire
  - University Hospital Coventry & Warwickshire, Coventry, Warwickshire
  - Wickersley Health Centre - Clifton Medical Centre, Rotherham

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] De Block C, Peleshok J, Wilding JPH, Kwan AYM, Rasouli N, Maldonado JM, Wysham C, Liu M, Aleppo G, Benneyworth BD. Post Hoc Analysis of SURPASS-1 to -5: Efficacy and Safety of Tirzepatide in Adults with Type 2 Diabetes are Independent of Baseline Characteristics. Diabetes Ther. 2025 Jan;16(1):43-71. doi: 10.1007/s13300-024-01660-0. Epub 2024 Nov 12. PMID 39531161
- [Derived] Osumili B, Fan L, Paik JS, Pantalone KM, Ranta K, Sapin H, Tofe S. Tirzepatide 5, 10 and 15 mg versus injectable semaglutide 0.5 mg for the treatment of type 2 diabetes: An adjusted indirect treatment comparison. Diabetes Res Clin Pract. 2024 Jun;212:111717. doi: 10.1016/j.diabres.2024.111717. Epub 2024 May 21. PMID 38777128
- [Derived] Boye KS, Sapin H, Dong W, Williamson S, Lee CJ, Thieu VT. Improved Glycaemic and Weight Management Are Associated with Better Quality of Life in People with Type 2 Diabetes Treated with Tirzepatide. Diabetes Ther. 2023 Nov;14(11):1867-1887. doi: 10.1007/s13300-023-01457-7. Epub 2023 Sep 5. PMID 37668888
- [Derived] Boye KS, Thieu VT, Sapin H, Lee CJ, Lando LF, Brown K, Bray R, Wiese RJ, Patel H, Rodriguez A, Yu M. Patient-Reported Outcomes in People with Type 2 Diabetes Receiving Tirzepatide in the SURPASS Clinical Trial Programme. Diabetes Ther. 2023 Nov;14(11):1833-1852. doi: 10.1007/s13300-023-01451-z. Epub 2023 Aug 1. PMID 37526908
- [Derived] Reitzel SB, Bogelund M, Basse A, Barszczewska O, Ren H. Semaglutide versus tirzepatide for people with type 2 diabetes: cost of glycemic control in Austria, the Netherlands, Lithuania, and the United Arab Emirates. Curr Med Res Opin. 2023 Aug;39(8):1055-1060. doi: 10.1080/03007995.2023.2231275. Epub 2023 Jul 10. PMID 37415503
- [Derived] Viljoen A, Pantalone KM, Galindo RJ, Cui X, Huh R, Hemmingway A, Fernandez Lando L, Patel H. Time to Reach Glycaemic and Body Weight Loss Thresholds with Tirzepatide in Patients with Type 2 Diabetes: A Pre-planned Exploratory Analysis of SURPASS-2 and SURPASS-3. Diabetes Ther. 2023 May;14(5):925-936. doi: 10.1007/s13300-023-01398-1. Epub 2023 Mar 31. PMID 37000390
- [Derived] Ten Doesschate T, van der Vaart TW, Debisarun PA, Taks E, Moorlag SJCFM, Paternotte N, Boersma WG, Kuiper VP, Roukens AHE, Rijnders BJA, Voss A, Veerman KM, Kerckhoffs APM, Oever JT, van Crevel R, van Nieuwkoop C, Lalmohamed A, van de Wijgert JHHM, Netea MG, Bonten MJM, van Werkhoven CH. Bacillus Calmette-Guerin vaccine to reduce healthcare worker absenteeism in COVID-19 pandemic, a randomized controlled trial. Clin Microbiol Infect. 2022 Sep;28(9):1278-1285. doi: 10.1016/j.cmi.2022.04.009. Epub 2022 Apr 28. PMID 35489606
- [Derived] Sattar N, McGuire DK, Pavo I, Weerakkody GJ, Nishiyama H, Wiese RJ, Zoungas S. Tirzepatide cardiovascular event risk assessment: a pre-specified meta-analysis. Nat Med. 2022 Mar;28(3):591-598. doi: 10.1038/s41591-022-01707-4. Epub 2022 Feb 24. PMID 35210595
- [Derived] Frias JP, Davies MJ, Rosenstock J, Perez Manghi FC, Fernandez Lando L, Bergman BK, Liu B, Cui X, Brown K; SURPASS-2 Investigators. Tirzepatide versus Semaglutide Once Weekly in Patients with Type 2 Diabetes. N Engl J Med. 2021 Aug 5;385(6):503-515. doi: 10.1056/NEJMoa2107519. Epub 2021 Jun 25. PMID 34170647
- See also: A Study of Tirzepatide (LY3298176) Versus Semaglutide Once Weekly as Add-on Therapy to Metformin in Participants With Type 2 Diabetes — https://trials.lillytrialguide.com/en-US/trial/4c6UpSKPWegDblIILD6NMM

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1 mg Semaglutide
Started | 471 | 469 | 470 | 469
Received at Least One Dose of Study Drug | 470 | 469 | 470 | 469
Completed | 452 | 442 | 446 | 443
Not Completed | 19 | 27 | 24 | 26
Not completed — Adverse Event | 1 | 4 | 1 | 3
Not completed — Death | 4 | 4 | 4 | 1
Not completed — Lost to Follow-up | 5 | 6 | 8 | 12
Not completed — Physician Decision | 0 | 2 | 0 | 4
Not completed — Pregnancy | 1 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Site terminated by Sponsor | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 7 | 8 | 4
Not completed — Other - as reported by the investigator | 1 | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- 5 mg Tirzepatide: 5 mg tirzepatide administered SC once a week.
- Total: Total of all reporting groups
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1 mg Semaglutide | Total
Number analyzed (Participants) | 470 | 469 | 470 | 469 | 1878
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (10.0) | 57.2 (10.5) | 55.9 (10.4) | 56.9 (10.8) | 56.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 265 | 231 | 256 | 244 | 996
  Male | 205 | 238 | 214 | 225 | 882
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 325 | 322 | 334 | 336 | 1317
  Not Hispanic or Latino | 145 | 147 | 136 | 133 | 561
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 53 | 53 | 57 | 45 | 208
  Asian | 6 | 11 | 5 | 3 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 2 | 3
  Black or African American | 28 | 21 | 15 | 15 | 79
  White | 382 | 376 | 392 | 401 | 1551
  More than one race | 1 | 8 | 0 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 158 | 160 | 161 | 161 | 640
  Australia | 12 | 11 | 12 | 11 | 46
  Brazil | 37 | 37 | 36 | 37 | 147
  Canada | 15 | 15 | 14 | 15 | 59
  Israel | 22 | 22 | 22 | 21 | 87
  Mexico | 89 | 87 | 88 | 88 | 352
  Puerto Rico | 6 | 4 | 6 | 3 | 19
  United Kingdom | 18 | 18 | 18 | 18 | 72
  United States | 113 | 115 | 113 | 115 | 456
Hemoglobin A1c [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 8.32 (1.08) | 8.30 (1.02) | 8.26 (1.00) | 8.25 (1.01) | 8.28 (1.03)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) (10 mg and 15 mg)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with Baseline + Pooled Country + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 40
Population: All participants who received at least one dose of study drug and had a baseline and at least 1 post-baseline HbA1c value, excluding patients who discontinued study drug due to inadvertent enrollment and data after initiating rescue antihyperglycemic medication or prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | 1 mg Semaglutide
Number analyzed (Participants) | 459 | 464 | 461
Percentage of HbA1c | -2.37 (0.048) | -2.46 (0.048) | -1.86 (0.048)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.51, 95% CI 2-sided [-0.64 to -0.38]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.60, 95% CI 2-sided [-0.73 to -0.47]

2. Secondary Outcome: Change From Baseline in HbA1c (5 mg)
Description: as for outcome 1
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 5 mg Tirzepatide | 1 mg Semaglutide
Number analyzed (Participants) | 461 | 461
Percentage of HbA1c | -2.09 (0.047) | -1.86 (0.048)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.23, 95% CI 2-sided [-0.36 to -0.10]

3. Secondary Outcome: Change From Baseline in Body Weight
Description: Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with Baseline + Pooled Country + Baseline HbA1c Group (<=8.5%, >8.5%) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 40
Population: All participants who received at least one dose of study drug and had a baseline and at least 1 post-baseline body weight value, excluding patients who discontinued study drug due to inadvertent enrollment and data after initiating rescue antihyperglycemic medication or prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: Kilograms (kg)
Groups:
- 1 mg Semaglutide: 1 mg of semaglutide administered SC once a week.
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1 mg Semaglutide
Number analyzed (Participants) | 461 | 459 | 464 | 462
Kilograms (kg) | -7.8 (0.33) | -10.3 (0.34) | -12.4 (0.34) | -6.2 (0.33)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.7, 95% CI 2-sided [-2.6 to -0.7]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -4.1, 95% CI 2-sided [-5.0 to -3.2]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -6.2, 95% CI 2-sided [-7.1 to -5.3]

4. Secondary Outcome: Percentage of Participants Achieving an HbA1c Target Value of <7%
Description: Hemoglobin A1c (HbA1c) is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1 mg Semaglutide
Number analyzed (Participants) | 461 | 459 | 464 | 461
Percentage of Participants | 85.47 | 88.89 | 92.24 | 81.13
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p = 0.023, Regression, Logistic; Odds Ratio (OR) = 1.54, 95% CI 2-sided [1.06 to 2.23]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.14, 95% CI 2-sided [1.44 to 3.17]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.03, 95% CI 2-sided [1.97 to 4.66]

5. Secondary Outcome: Change From Baseline in Fasting Serum Glucose (FSG)
Description: Fasting serum glucose (FSG) is a test to determine sugar levels in serum sample after an overnight fast. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with Baseline + Pooled Country + Baseline HbA1c Group (<=8.5%, >8.5%) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 40
Population: All participants who received at least one dose of study drug and had a baseline and at least 1 post-baseline FSG value, excluding patients who discontinued study drug due to inadvertent enrollment and data after initiating rescue antihyperglycemic medication or prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: milligram per Deciliter (mg/dL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1 mg Semaglutide
Number analyzed (Participants) | 461 | 458 | 464 | 459
milligram per Deciliter (mg/dL) | -56.0 (1.57) | -61.6 (1.60) | -63.4 (1.59) | -48.6 (1.58)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p = 0.001, Mixed Models Analysis; LS Mean Difference = -7.3, 95% CI 2-sided [-11.7 to -3.0]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -13.0, 95% CI 2-sided [-17.4 to -8.6]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -14.7, 95% CI 2-sided [-19.1 to -10.3]

6. Secondary Outcome: Mean Change From Baseline in Daily Average 7-Point Self-Monitored Blood Glucose (SMBG) Values
Description: The self-monitored plasma glucose (SMBG) data were collected at the following 7 time points: Morning Premeal - Fasting, Morning 2-hour Postmeal, Midday Premeal, Midday 2-hour Postmeal, Evening Premeal, Evening 2-hour Postmeal and Bedtime. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with Baseline + Pooled Country + Baseline HbA1c Group (<=8.5%, >8.5%) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 40
Population: All participants who received at least one dose of study drug and had a baseline and at least 1 post-baseline SMBG value, excluding patients who discontinued study drug due to inadvertent enrollment and data after initiating rescue antihyperglycemic medication or prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1 mg Semaglutide
Number analyzed (Participants) | 424 | 412 | 413 | 414
mg/dL | -65.4 (1.04) | -70.6 (1.05) | -74.3 (1.05) | -61.4 (1.04)

7. Secondary Outcome: Percentage of Participants Who Achieved Weight Loss ≥5%
Description: Percentage of Participants who Achieved Weight Loss ≥5%.
Time Frame: Week 40
Population: All participants who received at least one dose of study drug and had a baseline and at least 1 post-baseline weight loss, excluding patients who discontinued study drug due to inadvertent enrollment and data after initiating rescue antihyperglycemic medication or prematurely stopping study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1 mg Semaglutide
Number analyzed (Participants) | 461 | 459 | 464 | 462
Percentage of Participants | 68.55 | 82.35 | 86.21 | 58.44
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 1.58, 95% CI 2-sided [1.20 to 2.08]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.49, 95% CI 2-sided [2.57 to 4.75]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.60, 95% CI 2-sided [3.32 to 6.38]

8. Secondary Outcome: Diabetes Treatment Satisfaction as Measured by the Diabetes Treatment Satisfaction Questionnaire, Change Version (DTSQc) Hyperglycemia, Hypoglycemia and Total Score
Description: DTSQc, an 8-item questionnaire, assesses relative change in treatment satisfaction perceived frequency of hyperglycemia, and perceived frequency of hypoglycemia from baseline to week 40 or early termination. The questionnaire consists of 8 items, 6 of which (1 and 4 through 8) assess treatment satisfaction. Each item is rated on a 7-point Likert scale. The scores from the 6 treatment satisfaction items are summed to a Total Treatment Satisfaction Score, which ranges from -18 to 18 where the higher the score the greater the improvement in satisfaction with treatment. The lower the score the greater the deterioration in satisfaction with treatment. The hyperglycemia and hypoglycemia scores range from -3 to 3 where negative scores indicate fewer problems with blood glucose levels and positive scores indicate more problems than before. LS Mean was determined by ANCOVA with Baseline DTSQs + Pooled Country + Baseline HbA1c Group (<=8.5%, >8.5%) + Treatment (Type III sum of squares).
Time Frame: Baseline, Week 40
Population: All randomized participants who received at least one dose of study drug. Last observation carried forward (LOCF) endpoint only carries forward the last non-baseline observations before rescue therapy or stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1 mg Semaglutide
Number analyzed (Participants) | 419 | 399 | 398 | 412
Units on a Scale
  Hyperglycemia: number analyzed (Participants) | 418 | 399 | 398 | 411
  Hyperglycemia | -1.3 (0.10) | -1.4 (0.10) | -1.5 (0.10) | -1.1 (0.10)
  Hypoglycemia: number analyzed (Participants) | 416 | 398 | 398 | 412
  Hypoglycemia | -0.7 (0.10) | -0.7 (0.10) | -0.8 (0.10) | -0.7 (0.10)
  Total Score: number analyzed (Participants) | 419 | 399 | 398 | 411
  Total Score | 15.7 (0.18) | 15.6 (0.19) | 16.1 (0.19) | 15.8 (0.19)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs 1 mg Semaglutide; Hyperglycemia; Test type: Superiority; p = 0.084, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.50 to 0.03]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs 1 mg Semaglutide; Hyperglycemia; Test type: Superiority; p = 0.050, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.54 to 0.00]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs 1 mg Semaglutide; Hyperglycemia; Test type: Superiority; p = 0.005, ANCOVA; LS Mean Difference = -0.39, 95% CI 2-sided [-0.66 to -0.12]
Statistical Analysis 4: Comparison: 5 mg Tirzepatide vs 1 mg Semaglutide; Hypoglycemia; Test type: Superiority; p = 0.688, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.33 to 0.22]
Statistical Analysis 5: Comparison: 10 mg Tirzepatide vs 1 mg Semaglutide; Hypoglycemia; Test type: Superiority; p = 0.909, ANCOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.29 to 0.26]
Statistical Analysis 6: Comparison: 15 mg Tirzepatide vs 1 mg Semaglutide; Hypoglycemia; Test type: Superiority; p = 0.358, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.40 to 0.15]
Statistical Analysis 7: Comparison: 5 mg Tirzepatide vs 1 mg Semaglutide; Total Score; Test type: Superiority; p = 0.701, ANCOVA; LS Mean Difference = -0.10, 95% CI 2-sided [-0.62 to 0.41]
Statistical Analysis 8: Comparison: 10 mg Tirzepatide vs 1 mg Semaglutide; Total Score; Test type: Superiority; p = 0.341, ANCOVA; LS Mean Difference = -0.25, 95% CI 2-sided [-0.78 to 0.27]
Statistical Analysis 9: Comparison: 15 mg Tirzepatide vs 1 mg Semaglutide; Total Score; Test type: Superiority; p = 0.321, ANCOVA; LS Mean Difference = 0.26, 95% CI 2-sided [-0.26 to 0.79]

9. Secondary Outcome: Rate of Hypoglycemia With Blood Glucose <54 Milligram/Deciliter (mg/dL) [<3.0 Millimole/Liter (mmol/L)] or Severe Hypoglycemia
Description: The hypoglycemia events were defined by participant reported events with blood glucose <54mg/dL) (<3.0 mmol/L] or severe hypoglycemia. Severe hypoglycemia is defined as an episode with severe cognitive impairment requiring the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. These episodes may be associated with sufficient neuroglycopenia to induce seizure or coma. The rate of postbaseline hypoglycemia was estimated by negative binomial model: number of episodes = Pooled Country + Baseline HbA1c Group (<=8.5%, >8.5%) + Treatment.
Time Frame: Baseline through Safety Follow-Up (Up to Week 44)
Population: All randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Error); unit: Episodes/participant/365.25 days
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1 mg Semaglutide
Number analyzed (Participants) | 470 | 469 | 470 | 469
Episodes/participant/365.25 days | 0.0102 (0.00423) | 0.0046 (0.00488) | 0.0202 (0.00840) | 0.0046 (0.00340)

10. Secondary Outcome: Percentage of Participants Achieving an HbA1c Target Value of <5.7%
Description: Percentage of Participants Achieving an HbA1c Target Value of <5.7%.
Time Frame: Week 40
Population: All randomized participants who received at least one dose of study drug and had a baseline and at least 1 post-baseline HbA1c value, excluding patients discontinuing study drug due to inadvertent enrollment and data after initiating rescue antihyperglycemic medication or prematurely stopping study drug
Measure: Number; unit: Percentage of Participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1 mg Semaglutide
Number analyzed (Participants) | 461 | 459 | 464 | 461
Percentage of Participants | 29.28 | 44.66 | 50.86 | 19.74
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.86, 95% CI 2-sided [1.35 to 2.57]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.94, 95% CI 2-sided [2.88 to 5.39]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs 1 mg Semaglutide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.10, 95% CI 2-sided [3.73 to 6.97]

ADVERSE EVENTS:
Time Frame: Baseline, Safety follow-up (44 Weeks)
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- 5 mg Tirzepatide: 5 mg tirzepatide administered subcutaneously (SC) once a week.
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | 1 mg Semaglutide
All-Cause Mortality (participants affected / at risk) | 4/470 | 4/469 | 4/470 | 1/469
Serious Adverse Events (participants affected / at risk) | 33/470 | 25/469 | 27/470 | 13/469
Other Adverse Events (participants affected / at risk) | 170/470 | 187/469 | 202/470 | 172/469
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5 mg Tirzepatide (N=470) | 10 mg Tirzepatide (N=469) | 15 mg Tirzepatide (N=470) | 1 mg Semaglutide (N=469)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acromegaly (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epiploic appendagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Complicated appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) | 4 (4)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 1/205 (1) | 0/238 (0) | 0/214 (0) | 0/225 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suspected covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronavirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/265 (1) | 0/231 (0) | 0/256 (0) | 0/244 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified stage iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/265 (0) | 0/231 (0) | 1/256 (1) | 0/244 (0)
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/265 (1) | 0/231 (0) | 0/256 (0) | 0/244 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1/265 (1) | 0/231 (0) | 0/256 (0) | 0/244 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0/265 (0) | 0/231 (0) | 0/256 (0) | 1/244 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Tirzepatide (N=470) | 10 mg Tirzepatide (N=469) | 15 mg Tirzepatide (N=470) | 1 mg Semaglutide (N=469)
Abdominal pain (Gastrointestinal disorders) | 14 (16) | 20 (25) | 24 (30) | 24 (29)
Constipation (Gastrointestinal disorders) | 31 (35) | 21 (23) | 21 (23) | 27 (32)
Diarrhoea (Gastrointestinal disorders) | 62 (120) | 77 (98) | 65 (102) | 54 (68)
Dyspepsia (Gastrointestinal disorders) | 34 (46) | 29 (43) | 43 (51) | 31 (42)
Nausea (Gastrointestinal disorders) | 82 (110) | 90 (121) | 104 (136) | 84 (126)
Vomiting (Gastrointestinal disorders) | 27 (35) | 39 (54) | 46 (61) | 39 (53)
Decreased appetite (Metabolism and nutrition disorders) | 35 (38) | 34 (43) | 42 (51) | 25 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT03987919/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT03987919/SAP_001.pdf